CLINICAL TRIAL: NCT02658656
Title: CSP #2003 - Exoskeleton Assisted-Walking in Persons With SCI: Impact on Quality of Life
Brief Title: Powered Exoskeletons in Persons With SCI
Acronym: (PEPSCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003
Record Dates: First submitted 2016-01-06; First posted 2016-01-20 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injury
Keywords: Exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Exoskeleton + Standard of Care (SOC) (Active Comparator): Patient will receive exoskeletal-assisted walking device for in home use for 4 months
  Interventions: Device: ReWalk 6.0
- Standard of Care (SOC) (No Intervention): Patient will receive standard of care (wheelchair use)

INTERVENTIONS:
Device: ReWalk 6.0 — Exoskeletal Assisted Walking Device
  Arms: Exoskeleton + Standard of Care (SOC)

SUMMARY:
Background Veterans with spinal cord injury (SCI) have many adverse secondary medical and quality of life (QOL) changes as a result of immobilization. Veterans with SCI who have completed rehabilitation after injury and are unable to ambulate receive a wheelchair as standard of care (SOC) for mobility. Powered exoskeletons are a technology that has recently become available as an alternate form of mobility by providing an external framework for support and computer controlled motorized hip and knee joints to assist with over ground ambulation.

DETAILED DESCRIPTION:
Administrative hold due to COVID-19 pandemic.

Background Veterans with spinal cord injury (SCI) have many adverse secondary medical and quality of life (QOL) changes as a result of immobilization. Veterans with SCI who have completed rehabilitation after injury and are unable to ambulate receive a wheelchair as standard of care (SOC) for mobility. Powered exoskeletons are a technology that has recently become available as an alternate form of mobility by providing an external framework for support and computer controlled motorized hip and knee joints to assist with overground ambulation.

Research Questions (Objectives) Will Veterans with chronic SCI of six months duration, who are medically stable and who use a wheelchair as SOC plus an exoskeletal-assisted walking (EAW) device in their home and community environments have clinically meaningful net improvements in mental health, bladder, bowel, and pain patient-reported outcomes compared with those who use only the SOC? Additionally, will the use of an EAW device for four months in the homes and/or communities of the participants result in a reduction of total body fat mass? Study Design A two-group (Intervention and Control), randomized, clinical trial will be performed with a one-year feasibility component. The Intervention group will receive SOC plus EAW. The Control group will receive SOC only. The study will require seven years in total to complete and includes fifteen VA SCI Services as study sites. A feasibility phase will be employed using a staggered start by initially starting six sites, four sites starting one year later, and 5 other sites starting two years later. These initial six sites will be used to assess the start-up activities [hiring, training, equipment procurement, Central Institutional Review Board (CIRB) paperwork, etc.], the rate of recruitment, and any other issues that may be of value for the successful completion of the study. Lessons learned will be implemented for the remaining sites.

Relevance to VA In pilot studies conducted at the James J. Peters VA Medical Center, Bronx, NY, improvements in mental-emotional health, physical health and body composition were demonstrated by providing the participants the ability to walk for 4 to 6 hours per week over the course of three to five months. As of July 2014, a Class 2 designation was established by the Food and Drug Administration (FDA) for "powered exoskeletons". To date, one device (ReWalk ) has received FDA Class 2 approval for institutional and home use and is currently available by prescription. The Department of Veterans Affairs (DVA) is the largest single provider to persons with SCI in the USA, caring for about 26,000 of the 42,000 estimated Veterans with SCI. The VA presently lacks the infrastructure to support Veterans with SCI to train to use this device in order to make this technology available for the home/community use. A controlled research study would be anticipated to be the optimal manner to demonstrate the efficacy, amount of use and safety of a powered exoskeleton in the home and community environments; findings would be immediately transferable to clinical care.

Number of Research Participants (Sample Size) One hundred-sixty participants (80/group) will be randomized. Each of the 15 study sites will be expected to pre-screen 100 potential participants, screen 60 participants, to reach the target of 160 randomized over 15 sites.

Participating Sites Fifteen SCI Services will be selected on the basis of potential recruitment numbers (N=13,606 total Veterans with SCI in the sites' catchment areas and N=7,022 followed annually at these sites) and geographic location, to permit an even distribution across the country. The fifteen sites include: Boston, Richmond, St. Louis, Tampa, Milwaukee, Minneapolis, Dallas, Houston, Palo Alto, Long Beach, Augusta, San Antonio, Bronx, Cleveland, and Albuquerque. Of these fifteen sites, five are VA Cooperative Studies Program (CSP) Network of Dedicated Enrollment Sites (NODES).

Duration of Participant Intake (Study Duration) The CS #2003 study duration is projected to be a total of seven years: The initial six sites will have a start-up year, followed by participant enrollment/data collection during years 1-4, and continued data collection/closeout during year 5, for a total of six years. The next four sites will begin the start-up year one year after the first six sites and follow the same enrollment, data collection and closeout schedule over the next five years. The next five sites will begin start-up one year after the four sites and follow the same enrollment, data collection and closeout schedule. All fifteen sites will be closed out after six years, and there is an additional year for the Coordinating Center and Chairperson's Office to complete data analysis and manuscript writing, thus the study total time is seven years. Participants in both groups will be asked to commit 33 weeks to this study. Participants in the Control arm will be offered an additional 8 weeks to receive EAW training in the medical centers, without outcome data being collected.

Treatment (follow-up) The intervention being tested is four months of home and/or community use of a powered exoskeleton.

Definition of Participant Samples (Study Population) One-hundred sixty male or female Veterans or military members with chronic SCI, six months duration, 18 years of age, functional use of their hands, medically stable, and wheelchair users for indoor and outdoor mobility, will be eligible for screening. All potential participants will be Veterans or military members with SCI. Study participants will generally be outpatients with the exception of those inpatients who meet the eligibility criteria, and who are approved by the Site Investigator (e.g., some inpatients may have been admitted for a wheelchair fitting or another non-medical reason). Non-veterans with SCI will not be eligible.

Treatment Arms All participants will receive four months of treatment, randomized into two arms: SOC plus EAW or SOC only.

Endpoints Primary outcome one will be the Mental Component Summary of the Veterans Rand-36 (MCS/VR-36). Primary outcome two will be the sum T-score of the SCI-QOL bladder management difficulties, bowel management difficulties and pain interference item banks. The major secondary outcome will be total body fat mass. The two primary and the major secondary outcomes will be analyzed as the proportion of participants in each group who achieved a clinically meaningful change in score. The endpoint will be success or failure for these outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans or active duty military personnel who are at least 18 years of age;
2. Traumatic or non-traumatic SCI 6 months duration of SCI;
3. Wheelchair-user for indoor and outdoor mobility;
4. Anthropometric compatibility with the device:

   1. Weight <220 lb. (100 kg),
   2. Thigh length between 14 and 19 in (36 and 48 cm),
   3. Shank length between 17 and 22 in (43 and 55 cm);
5. Able to hold the crutches in hands without modifications;
6. Able to have a companion who can attend approximately one-third of the training sessions who will assist them at home and in the community; and
7. Able to provide informed consent.

Exclusion Criteria:

1. Diagnosis of neurological injury other than SCI;
2. Progressive condition that would be expected to result in changing neurological status;
3. Severe concurrent medical disease, illness or condition judged to be contraindicated by the Site Physician;
4. Unhealed or unstable traumatic or high impact lower extremity fracture (definition below) of any duration that is in the clinical judgement of the study physician to be exclusionary for standing and walking;
5. Knee BMD < 0.60 gm/cm2;
6. Total hip BMD T-scores < -3.5;
7. Fragility, minimal trauma or low impact fracture of the lower extremity since spinal cord injury (definition below);
8. Untreatable severe spasticity judged to be contraindicated by the Site Physician;
9. Flexion contracture > 15 degrees at the hip and/or > 10 degrees at the knee;
10. Limitations in ankle range of motion that cannot be adapted with an orthotic device (plantar flexion > 00);
11. Untreated or uncontrolled hypertension (systolic blood pressure >140 mmHg; diastolic blood pressure >90 mmHg);
12. Unresolved orthostatic hypotension (systolic blood pressure <90 mmHg; diastolic blood pressure <60 mmHg) as judged to be contraindicated by the Site Physician;
13. Current pressure ulcer of the arms, trunk, pelvic area, or lower extremities;
14. Psychopathology documentation in the medical record or history that may conflict with study objectives; and/or
15. Pregnancy or women who plan to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Spungen, EdD, Study Chair — James J. Peters Veterans Affairs Medical Center
Locations (15):
- United States (15):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared.

REFERENCES:
- [Result] Spungen AM, Dematt EJ, Biswas K, Jones KM, Mi Z, Snodgrass AJ, Morin K, Asselin PK, Cirnigliaro CM, Kirshblum S, Gorman PH, Goetz LL, Stenson K, White KT, Hon A, Sabharwal S, Kiratli BJ, Ota D, Bennett B, Berman JE, Castillo D, Lee KK, Eddy BW, Henzel MK, Trbovich M, Holmes SA, Skelton F, Priebe M, Kornfeld SL, Huang GD, Bauman WA. Exoskeletal-Assisted Walking in Veterans With Paralysis: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2431501. doi: 10.1001/jamanetworkopen.2024.31501. PMID 39230903

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Patient will receive standard of care (wheelchair use)
- Screen Failures: Consented participants who failed screening and were not randomized.
Period: Screening
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care | Screen Failures
Started | 78 | 83 | 263
Completed | 78 | 83 | 0
Not Completed | 0 | 0 | 263
Not completed — Failed eligibility criteria | 0 | 0 | 263
Period: Randomization
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care | Screen Failures
Started | 78 | 83 | 0
Completed | 45 | 57 | 0
Not Completed | 33 | 26 | 0
Not completed — Withdrawal by Subject | 8 | 7 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Administrative Termination | 3 | 1 | 0
Not completed — Administrative Termination due to COVID-19 Restrictions | 13 | 15 | 0
Not completed — Failed Exoskeletal-assisted walking (EAW) Advanced Skills Test | 2 | 0 | 0
Not completed — Not eligible for Randomization | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exoskeleton + SOC: Patient will receive exoskeletal-assisted walking device for in home use for 4 months
  ReWalk 6.0: Exoskeletal Assisted Walking Device
- Total: Total of all reporting groups
Arm/Group | Exoskeleton + SOC | Standard of Care | Total
Number analyzed (Participants) | 78 | 83 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.61) | 46.2 (13.27) | 46.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 72 | 79 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 19 | 27
  Not Hispanic or Latino | 66 | 63 | 129
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 55 | 54 | 109
  More than one race | 6 | 13 | 19
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 83 | 161
Mental Health Component Summary (MCS) of the Veterans Rand-36 (VR-36) [Mean (Standard Deviation); unit: units on a scale] — The Mental Health Component Summary (MCS) of the VR-36 measures the vitality, social functioning, role-emotional, and mental health of the participant. Possible range of the MCS is 0 to 100, with a higher score indicating higher mental wellbeing.
  units on a scale | 60.6 (10.85) | 59.2 (11.71) | 59.9 (11.29)
SCI-QOL Physical Medical Health Domain [Mean (Standard Deviation); unit: units on a scale] — The sum T-score for the SCI-QOL Physical Medical Health domain (three item banks of Bladder Management Difficulties, Bowel Management Difficulties, and Pain Interference). Possible score range is 110 to 253, with a lower score indicating better physical medical wellbeing.
  units on a scale | 153 (21.11) | 153 (23.93) | 153 (22.54)

OUTCOME MEASURES:

1. Primary Outcome: Improvement on the MCS in All Randomized Participants
Description: Number of randomized participants with a greater than or equal to 4 point change on the Mental Health Component Summary (MCS) of the Veterans Rand-36 (VR-36) from Baseline Assessment to 4 Months Post Intervention. Possible range of the MCS is 0 to 100, with a higher score indicating higher mental wellbeing.
Time Frame: Change from Baseline Assessment to 4 Months Post Intervention
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + SOC | Standard of Care
Number analyzed (Participants) | 78 | 83
Participants | 12 | 14
Statistical Analysis 1: Comparison: Exoskeleton + SOC vs Standard of Care; Test type: Superiority; p = 0.798, Chi-squared; Risk Ratio (RR) = 0.91, 95% CI 2-sided [.45 to 1.85]

2. Primary Outcome: Improvement on the SCI-QOL Physical Medical Health Domain in All Randomized Participants
Description: Number of randomized participants with a greater than or equal to 10 percent decrease on the SCI-QOL Physical Medical Health Domain (PMH) from Baseline Assessment to 4 Months Post Intervention. The PMH score is a sum of the SCI-QOL scores from the Bladder Management Difficulties, Bowel Management Difficulties, and Pain Interference item banks. Possible range of the PMH score is 110 to 253, with a lower score indicating better physical medical wellbeing.
Time Frame: Change from Baseline Assessment to 4 Months Post Intervention
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + SOC | Standard of Care
Number analyzed (Participants) | 78 | 83
Participants | 10 | 11
Statistical Analysis 1: Comparison: Exoskeleton + SOC vs Standard of Care; Test type: Superiority; p = 0.935, Chi-squared; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.44 to 2.15]

3. Secondary Outcome: Total Body Fat Loss in All Randomized Participants
Description: Number of randomized participants with a greater than or equal to 1kg of total body fat loss from Baseline Assessment to 4 Months Post Intervention
Time Frame: 4 months post intervention
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 78 | 83
Participants | 14 | 16
Statistical Analysis 1: Comparison: Exoskeleton + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority; p = 0.829, Chi-squared; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.49 to 1.79]

4. Secondary Outcome: Improvement on the Mental Health Component Summary (MCS) in Participants Who Completed the 4 Month Intervention Phase.
Description: Number of participants, out of those who completed the 4 month intervention phase, with a greater than or equal to 4 point increase on the Mental Health Component Summary (MCS) of the Veterans Rand-36 (VR-36) from Baseline Assessment to 4 Months Post Intervention. Possible range of the MCS is 0 to 100, with a higher score indicating higher mental wellbeing.
Time Frame: 4 months post intervention
Population: Participants who completed the 4 month intervention phase
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 57
Participants | 12 | 14
Statistical Analysis 1: Comparison: Exoskeleton + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority; p = 0.809, Chi-squared; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.56 to 2.11]

5. Secondary Outcome: Improvement on the SCI-QOL Physical Medical Health Domain in Participants Who Completed the 4 Month Intervention Phase.
Description: Number of participants, out of those who completed the 4 month intervention phase, with a greater than or equal to 10 percent improvement (decrease) on the Spinal Cord Injury Quality of Life (SCI-QOL) Physical Medical Health Domain (PMH) from Baseline Assessment to 4 Months Post Intervention. The PMH score is a sum of the SCI-QOL scores from the Bladder Management Difficulties, Bowel Management Difficulties, and Pain Interference item banks. Possible range of the PMH score is 110 to 253, with a lower score indicating better physical medical wellbeing.
Time Frame: 4 months post intervention
Population: Participants that completed the 4 month intervention phase
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 57
Participants | 10 | 11
Statistical Analysis 1: Comparison: Exoskeleton + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority; p = 0.717, Chi-squared; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.54 to 2.47]

6. Secondary Outcome: Total Body Fat Loss in Participants Who Completed the 4 Month Intervention Phase.
Description: Number of participants, out of those who completed the 4 month intervention phase, with a greater than or equal to 1kg of total body fat loss from Baseline Assessment to 4 Months Post Intervention
Time Frame: 4 months post intervention
Population: participants who completed the 4 month intervention phase
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 57
Participants | 14 | 16
Statistical Analysis 1: Comparison: Exoskeleton + Standard of Care (SOC) vs Standard of Care (SOC); Test type: Superiority; p = 0.738, Chi-squared; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.61 to 2.02]

7. Secondary Outcome: Change in Mental Health Component Summary (MCS)
Description: Mean difference score in the Mental Health Component Summary (MCS) of the Veterans Rand-36 (VR-36) from baseline to post training/orientation, two months post intervention, and 4 months post intervention. Possible range of the MCS is 0 to 100, with a higher score indicating higher mental wellbeing.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a Mental Health Component Summary (MCS) score at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 73
score on a scale
  Post training/orientation: number analyzed (Participants) | 54 | 67
  Post training/orientation | 1.7 (9.57) | -0.3 (7.32)
  2 month post intervention: number analyzed (Participants) | 48 | 59
  2 month post intervention | 1.0 (8.04) | -1.0 (8.42)
  4 month post intervention: number analyzed (Participants) | 45 | 56
  4 month post intervention | -0.1 (10.40) | -1.8 (10.38)

8. Secondary Outcome: Change in SCI-QOL Physical Medical Health Domain
Description: Mean difference score in the SCI-QOL Physical Medical Health Domain from baseline to post training/orientation, two months post intervention, and 4 months post intervention. The PMH score is a sum of the SCI-QOL scores from the Bladder Management Difficulties, Bowel Management Difficulties, and Pain Interference item banks. Possible range of the PMH score is 110 to 253, with a lower score indicating better physical medical wellbeing.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a PMH score at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 73
score on a scale
  Post training/orientation: number analyzed (Participants) | 54 | 67
  Post training/orientation | -4.4 (17.60) | -0.5 (16.59)
  2 month post intervention: number analyzed (Participants) | 47 | 58
  2 month post intervention | -5.9 (15.56) | -1.7 (17.73)
  4 month post intervention: number analyzed (Participants) | 43 | 57
  4 month post intervention | -6.9 (17.71) | -1.5 (19.99)

9. Secondary Outcome: Change in Total Body Fat
Description: Change in total body fat from baseline to post training/orientation, two months post intervention, and 4 months post intervention
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a total body fat measurement at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 73
kilograms
  Post training/orientation: number analyzed (Participants) | 54 | 65
  Post training/orientation | 0.2 (2.01) | 0.3 (1.82)
  2 month post intervention: number analyzed (Participants) | 47 | 57
  2 month post intervention | 0.4 (3.13) | 0.1 (2.84)
  4 month post intervention: number analyzed (Participants) | 45 | 55
  4 month post intervention | 0.1 (3.75) | 0.1 (3.59)

10. Secondary Outcome: Change in SCI-QOL Social Participation Domain
Description: Mean difference score in the SCI-QOL Social Health Domain from baseline to post training/orientation, two months post intervention, and 4 months post intervention. The Social Health Domain score is a sum of the SCI-QOL scores from the ability to participate in social roles and activities, satisfaction with social roles and activities, and independence item banks. Possible range of the Social Health Domain score is 78 to 191, with a higher score indicating higher social health.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a Social Health Domain score at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 52 | 74
score on a scale
  post training/orientation: number analyzed (Participants) | 52 | 68
  post training/orientation | 1.9 (14.74) | -2.0 (13.58)
  2 month post intervention: number analyzed (Participants) | 46 | 59
  2 month post intervention | -0.2 (17.13) | -2.2 (13.45)
  4 month post intervention: number analyzed (Participants) | 43 | 57
  4 month post intervention | 4.1 (15.00) | -3.0 (16.59)

11. Secondary Outcome: Change in SCI-QOL Positive Emotional Constraints
Description: Mean difference score in the SCI-QOL Positive Emotional Constraints from baseline to post training/orientation, two months post intervention, and 4 months post intervention. The Positive Emotional Constraints score is a sum of the SCI-QOL scores from the positive affect and well being, self-esteem, and resilience item banks. Possible range of the Positive Emotional Constraints score is 63 to 199, with a higher score indicating better emotional wellbeing.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a score on the SCI-QOL Positive Emotional Constraints at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 73
score on a scale
  Post Training/Orientation: number analyzed (Participants) | 54 | 67
  Post Training/Orientation | 0.1 (17.72) | -2.3 (16.87)
  2 months post intervention: number analyzed (Participants) | 48 | 59
  2 months post intervention | 1.7 (16.28) | -1.8 (16.71)
  4 months post intervention: number analyzed (Participants) | 45 | 56
  4 months post intervention | 2.6 (14.99) | -3.2 (20.63)

12. Secondary Outcome: Change in SCI-QOL Negative Emotional Constraints
Description: Mean difference score in the SCI-QOL Negative Emotional Constraints from baseline to post training/orientation, two months post intervention, and 4 months post intervention. The Negative Emotional Constraints score is a sum of the SCI-QOL scores from the anxiety, depression, grief-loss, trauma, and stigma item banks. Possible range of the Negative Emotional Constraints score is 182 to 405, with a lower score indicating better emotional wellbeing.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a score on SCI-QOL Negative Emotional Constraints at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 74
Score on a scale
  post training/orientation: number analyzed (Participants) | 54 | 68
  post training/orientation | -6.5 (25.20) | 3.6 (22.42)
  2 months post intervention: number analyzed (Participants) | 48 | 60
  2 months post intervention | -8.4 (21.83) | 1.1 (22.05)
  4 months post intervention: number analyzed (Participants) | 44 | 57
  4 months post intervention | -8.6 (22.34) | 1.5 (26.91)

13. Secondary Outcome: Change in SCI Functional Index (FI)
Description: Mean difference score in the SCI Functional Index (FI) from baseline to post training/orientation, two months post intervention, and 4 months post intervention. The SCI Function Index for physical function is a sum of the basic mobility, ambulation, fine motor, self-care, and wheelchair mobility item banks. Possible range of the SCI Functional Index is 188 to 408, with a higher score indicating better physical function.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a score on the SCI FI at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 21 | 23
score on a scale
  Post Training/Orientation: number analyzed (Participants) | 18 | 19
  Post Training/Orientation | 5.4 (20.97) | -5.8 (11.63)
  Two months post intervention: number analyzed (Participants) | 16 | 19
  Two months post intervention | 7.3 (16.00) | -4.5 (12.99)
  4 months post intervention: number analyzed (Participants) | 17 | 17
  4 months post intervention | 3.8 (16.36) | -8.6 (20.60)

14. Secondary Outcome: Change in Sleep Disturbance
Description: Mean difference T-score of the Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance from baseline to post training/orientation, two months post intervention, and 4 months post intervention. Possible range of the PROMIS is 28.9 to 76.5, with a higher score indicating more sleep disturbance.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized with a score on the PROMIS Sleep Disturbance score at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 74
Score on a scale
  Post Training/Orientation: number analyzed (Participants) | 54 | 68
  Post Training/Orientation | -1.8 (8.83) | 2.1 (7.57)
  2 months post intervention: number analyzed (Participants) | 48 | 59
  2 months post intervention | -2.1 (8.75) | 1.6 (7.50)
  4 months post intervention: number analyzed (Participants) | 45 | 57
  4 months post intervention | -0.3 (9.91) | 1.3 (7.58)

15. Secondary Outcome: Change in Participant Impression of Severity
Description: Mean difference in the participant impression of severity of spinal cord injury from the Global Impression of Change Scale from baseline to post training/orientation, two months post intervention, and 4 months post intervention. Possible range of the participant impression of severity is 1 to 7, with a higher score indicating worse impression of severity of spinal cord injury.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with an impression of severity score on the Global Impression of Change Scale at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 73
score on a scale
  Post Training/Orientation: number analyzed (Participants) | 54 | 66
  Post Training/Orientation | -0.2 (1.10) | 0.4 (1.06)
  2 months post intervention: number analyzed (Participants) | 47 | 58
  2 months post intervention | 0.0 (1.01) | 0.3 (1.13)
  4 months post intervention: number analyzed (Participants) | 44 | 56
  4 months post intervention | -0.1 (1.17) | 0.3 (1.16)

16. Secondary Outcome: Change in Companion Impression of Severity
Description: Mean difference in the companion impression of severity of spinal cord injury from the Global Impression of Change Scale from baseline to post training/orientation, two months post intervention, and 4 months post intervention. Possible range of the companion impression of severity is 1 to 7, with a higher score indicating worse impression of severity of spinal cord injury.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a companion impression of severity score on the Global Impression of Change Scale at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 52 | 72
score on a scale
  Post Training/Orientation: number analyzed (Participants) | 51 | 63
  Post Training/Orientation | 0.0 (1.30) | 0.0 (1.13)
  Two months post intervention: number analyzed (Participants) | 45 | 56
  Two months post intervention | 0.2 (1.55) | 0.3 (1.48)
  4 months post intervention: number analyzed (Participants) | 41 | 51
  4 months post intervention | 0.2 (1.28) | 0.3 (1.13)

17. Secondary Outcome: Bowel Evacuation Time
Description: Time spent to have a bowel movement per bowel day, over 7 days. Responses were collected using a 5-point likert scale with the following options: 5 to 15 minutes; 15 to 30 minutes; 30 to 60 minutes; 1 to 3 hours; more than 3 hours.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 56
Participants
  5 to 15 minutes | 14 | 8
  15 to 30 minutes | 10 | 14
  30 to 60 minutes | 10 | 22
  1 to 3 hours | 10 | 11
  More than 3 hours | 1 | 1

18. Secondary Outcome: Frequency of Bowel Evacuation Episodes
Description: Frequency of bowel movements over 7 days. Responses were collected using a 5-point Likert scale with the following options: 7 times or more; 5 to 6 times; 3 to 4 times; 1 to 2 times; none.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 55
Participants
  7 times or more | 18 | 23
  5-6 times | 7 | 9
  3-4 times | 16 | 16
  1-2 times | 4 | 6
  None | 0 | 1

19. Secondary Outcome: Manual/Digit Stimulation for Bowel Movements
Description: Needed manual/digit stimulation for bowel movements over 7 days. Responses were collected using a 5-point Likert scale with the following options: none/never; only once; a few times; most times; every time.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 56
Participants
  None/never | 11 | 11
  Only once | 1 | 3
  A few times | 5 | 6
  Most times | 4 | 4
  Every time | 24 | 32

20. Secondary Outcome: Oral Medications for Bowel Movements
Description: Required oral medications to help with bowel movements over 7 days. Responses were collected using a 5-point Likert scale with the following options: none/never; only once; a few times; most times; every time.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 56
Participants
  None/never | 22 | 33
  Only once | 1 | 3
  A few times | 6 | 2
  Most times | 3 | 2
  Every time | 13 | 16

21. Secondary Outcome: Enemas or Irrigations for Bowel Movements
Description: Required enemas or irrigations to help with bowel movements over 7 days. Responses were collected using a 5-point Likert scale with the following options: none/never; only once; a few times; most times; every time.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 56
Participants
  None/never | 30 | 33
  Only once | 1 | 4
  A few times | 4 | 4
  Most times | 1 | 2
  Every time | 9 | 13

22. Secondary Outcome: Bowel Control
Description: Bowel accidents over 7 days. Responses were collected using a 5-point Likert scale with the following options: no leakage or accidents; leakage or an accident 1-2 times; leakage or an accident 3-4 times; leakage or an accident 5-6 times; leakage or an accident 7 or more times.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 45 | 56
Participants
  No leakage or accidents | 31 | 43
  Leakage or an accident 1-2 times | 12 | 11
  Leakage or an accident 3-4 times | 2 | 1
  Leakage or an accident 5-6 times | 0 | 0
  Leakage or an accident 7 or more times | 0 | 1

23. Secondary Outcome: Stool Consistency
Description: Stool consistency by the Bristol Stool Scale over 7 days. The Bristol Stool Scale classifies stools into seven groups: separate hard lumps; sausage-shaped, but lumpy; like sausage, cracks on surface; like a snake, smooth and soft; soft blobs (passed easily); fluffy pieces, a mush stool; watery, entirely liquid.
Time Frame: 4 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 42 | 55
Participants
  Separate hard lumps | 1 | 4
  Sausage-shaped, but lumpy | 5 | 10
  Like sausage, cracks on surface | 13 | 14
  Like a snake, smooth and soft | 11 | 21
  Soft blobs (passed easily) | 5 | 2
  Fluffy pieces, a mush stool | 7 | 2
  Watery, entirely liquid | 0 | 2

24. Secondary Outcome: Change in Abdominal Fat Mass
Description: Change in visceral adipose tissue mass measured from bone density scan, in grams, from baseline to post training/orientation, two months post intervention, and 4 months post intervention
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a bone density scan at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 54 | 73
grams
  Post Training/Orientation: number analyzed (Participants) | 54 | 64
  Post Training/Orientation | 57 (269.4) | 30 (247.8)
  Two months post intervention: number analyzed (Participants) | 47 | 57
  Two months post intervention | 93 (351.6) | 2 (247.4)
  4 months post intervention: number analyzed (Participants) | 45 | 55
  4 months post intervention | 67 (360.2) | 21 (273.4)

25. Secondary Outcome: Change in High Density Lipoprotein Cholesterol
Description: Change in high density lipoprotein cholesterol, in milligrams per deciliter (mg/dL), from baseline to post training/orientation, two months post intervention, and 4 months post intervention
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a high density lipoprotein cholesterol lab value at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 49 | 66
mg/dL
  Post Training/Orientation: number analyzed (Participants) | 47 | 59
  Post Training/Orientation | 0.8 (6.55) | -0.6 (8.66)
  Two Months post intervention: number analyzed (Participants) | 42 | 51
  Two Months post intervention | 1.3 (6.42) | 0.2 (8.11)
  4 months post intervention: number analyzed (Participants) | 37 | 48
  4 months post intervention | 0.7 (7.3) | -0.3 (7.5)

26. Secondary Outcome: Change in Low Density Lipoprotein Cholesterol
Description: Change in low density lipoprotein cholesterol, in milligrams per deciliter (mg/dL), from baseline to post training/orientation, two months post intervention, and 4 months post intervention
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a low density lipoprotein cholesterol lab value at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 48 | 65
mg/dL
  Post training/Orientation: number analyzed (Participants) | 46 | 59
  Post training/Orientation | -2.9 (24.26) | 1.2 (28.49)
  Two months post intervention: number analyzed (Participants) | 40 | 51
  Two months post intervention | -0.6 (21.15) | -0.7 (21.13)
  4 months post intervention: number analyzed (Participants) | 35 | 47
  4 months post intervention | -2.4 (20.77) | 1.8 (23.97)

27. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol, in milligrams per deciliter (mg/dL), from baseline to post training/orientation, two months post intervention, and 4 months post intervention
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a total cholesterol lab value at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 49 | 66
mg/dL
  Post Training/Orientation: number analyzed (Participants) | 47 | 59
  Post Training/Orientation | 2.9 (32.44) | 0.0 (31.42)
  Two months post intervention: number analyzed (Participants) | 42 | 51
  Two months post intervention | 2.6 (31.93) | 1.4 (26.08)
  4 Months post intervention: number analyzed (Participants) | 37 | 48
  4 Months post intervention | 4.8 (36.71) | 1.1 (29.65)

28. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides, in milligrams per deciliter (mg/dL), from baseline to post training/orientation, two months post intervention, and 4 months post intervention
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with a triglycerides lab value at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 49 | 66
mg/dL
  Post Training/Orientation: number analyzed (Participants) | 47 | 59
  Post Training/Orientation | 3.9 (61.78) | 4.0 (57.37)
  Two months post intervention: number analyzed (Participants) | 42 | 51
  Two months post intervention | 3.0 (68.36) | 9.5 (68.17)
  4 months post intervention: number analyzed (Participants) | 37 | 48
  4 months post intervention | 14.9 (104.2) | -2.3 (61.12)

29. Secondary Outcome: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Description: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), from baseline to post training/orientation, two months post intervention, and 4 months post intervention. HOMA-IR= Fasting insulin (mIU/ml) x Fasting glucose (mg/dl) / 405.
Time Frame: post training/orientation, two months post intervention, and 4 months post intervention.
Population: Randomized participants with fasting insulin and fasting glucose lab values at baseline and at least one of the following time points: post training/orientation, two months post intervention, or 4 months post intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exoskeleton + Standard of Care (SOC) | Standard of Care (SOC)
Number analyzed (Participants) | 51 | 65
units on a scale
  Post Training/Orientation: number analyzed (Participants) | 50 | 59
  Post Training/Orientation | 1.1 (3.94) | 0.1 (2.68)
  Two months post intervention: number analyzed (Participants) | 43 | 47
  Two months post intervention | 2.3 (11.4) | 0.1 (4.27)
  4 months post intervention: number analyzed (Participants) | 39 | 47
  4 months post intervention | 1.7 (8.11) | 0.3 (3.7)

ADVERSE EVENTS:
Time Frame: From consent to 4 month post intervention.
Description: Events reported in the not randomized column were events that occurred prior to randomization. Events that occurred after randomization are reported under the respective treatment group.
Groups:
- Prior to Randomization: Consented patients prior to randomization
Arm/Group | Exoskeleton + SOC | Standard of Care | Prior to Randomization
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/83 | 2/424
Serious Adverse Events (participants affected / at risk) | 11/78 | 14/83 | 27/424
Other Adverse Events (participants affected / at risk) | 54/78 | 44/83 | 86/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exoskeleton + SOC (N=78) | Standard of Care (N=83) | Prior to Randomization (N=424)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 3 (5) | 6 (6)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Drug use disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Botulinum toxin injection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Heart valve operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (3) | 4 (11) | 6 (7)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Penile prosthesis insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exoskeleton + SOC (N=78) | Standard of Care (N=83) | Prior to Randomization (N=424)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syringomyelia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0)
Medical device site bruise (General disorders) | 2 (5) | 0 (0) | 9 (11)
Medical device site erythema (General disorders) | 2 (2) | 0 (0) | 1 (3)
Medical device site haematoma (General disorders) | 1 (1) | 0 (0) | 1 (1)
Medical device site injury (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 12 (15) | 16 (23) | 15 (18)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Autonomic dysreflexia (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 4 (4)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (5) | 3 (3) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 17 (20) | 6 (14) | 7 (7)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Nail avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 7 (7) | 4 (6) | 4 (5)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 4 (4) | 2 (3) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen consumption increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Scan (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 4 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal atrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (5) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Apicectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Botulinum toxin injection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Breast conserving surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Elective surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (3) | 4 (7) | 5 (5)
Incisional hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02658656/Prot_SAP_000.pdf